CLINICAL TRIAL: NCT06715306
Title: Intravenous Versus Oral Treatment of the Main Acute Infections in Emergency Departments
Brief Title: Intravenous Versus Oral Treatment of the Main Acute Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHS-ED-1-2024
Record Dates: First submitted 2024-11-05; First posted 2024-12-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections; Cellulitis
Keywords: Oral antibiotic therapy; intravenous antibiotic therapy; intravenous-to-oral-switch
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections; Cellulitis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard intravenous treatment in accordance with local or national procedures
- Oral treatment (Active Comparator): Oral treatment
  Interventions: Other: Oral treatment

INTERVENTIONS:
Other: Oral treatment — Patients randomized to oral treatment will commence the oral treatment immediately. The oral treatment is based on specially developed treatment suggestions developed by microbiologists and specialists in infectious diseases from the participating regions, and in respect with local treatment guidelines (detailed described in the protocol).
  Arms: Oral treatment

SUMMARY:
Patients admitted to the hospital with acute infections are often treated with intravenous (IV) antibiotics. Around 70% of these infections fall into three categories: respiratory tract infections, urinary tract infections, and cellulitis. A Danish study found that 76% of patients admitted with suspected community-acquired pneumonia and treated with antibiotics received them intravenously. Based on an extrapolated estimate from an unpublished local survey, approximately 50,000 patients in Denmark are admitted each year for infections and treated with IV antibiotics. The average hospital stay for these patients is 5.9 days, resulting in a total of 295,000 hospital days annually, accounting for about 7% of total hospital admissions in Denmark. This represents an annual cost of 2.3 billion DKK. While some patients need hospitalization due to their overall health or other serious conditions, others remain hospitalized primarily to receive IV antibiotics.

Expanding the use of oral antibiotics in emergency departments should be pursued only if it can demonstrate comparable efficacy and safety to IV administration. Therefore this study will investigate the efficiency of primarily oral antibiotics in acutely admitted patients with proven or suspected infections. Additionally, the investigators will evaluate the safety of oral regimen for these patients.

DETAILED DESCRIPTION:
Patients admitted to the hospital with infections are often treated with intravenous antibiotics. The rationale for using intravenous antibiotics includes eliminating the risk of reduced absorption, achieving higher serum concentrations, and the fact that many broad-spectrum antibiotics (such as cephalosporins and carbapenems) are not available in oral form. However, intravenous antibiotics also have drawbacks, such as the risk of catheter-related infections, challenges in home-based treatment, and difficulty switching to oral antibiotics unless microbiological results are definitively positive. Prolonged hospital stays associated with intravenous antibiotic treatment lead to economic burdens, increased risk of hospital-acquired infections, and significant functional decline, especially in older patients.

In recent decades, many studies have explored the possibility of fully or partially replacing intravenous antibiotics with oral antibiotics for certain infections.

In this study, the investigators will examine the safety and efficacy of primarily oral antibiotic regimens in patients with confirmed or suspected infections admitted to the emergency department. The study is an open-label, prospective, randomized controlled trial. Participants will be randomly assigned to receive either standard intravenous antibiotic treatment according to Danish guidelines or oral antibiotic treatment based on tailored recommendations developed by microbiologists and infectious disease specialists at participating sites, in accordance with local guidelines.

The study has two primary outcomes: 1) Efficacy-measured as the number of days alive outside the hospital within 30 days after randomization, and 2) Safety-measured by mortality or the need for vasopressors within 30 days after randomization. A total of 4,000 patients will be needed to address both primary outcomes.

Aim: The trial aims to investigate the safety and efficacy of oral antibiotic administration compared to intravenous antibiotic administration in patients referred to the emergency department with suspected or diagnosed bacterial pneumonia, urinary tract infection and cellulitis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected respiratory tract infection, urinary tract infection, or cellulitis by the attending physician
* Planned or initiated intravenous antibiotic treatment

Exclusion Criteria:

* if received more than two doses of intravenous antibiotics;
* systolic blood pressure <90 mmHg;
* nausea and/or vomiting in more than one short-term instance during the last 2 days;
* suspected significantly reduced gastrointestinal absorption;
* confirmed plasma-lactate > 2;
* pregnant or nursing;
* unable to give informed consent;
* severe immunodeficiency;
* urgent vital treatment needed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2028-01-06 (Estimated)

PRIMARY OUTCOMES:
Days alive outside hospital (Efficacy) | From randomization date to 30 days
  The number of days the patients are alive outside hospital within 30 days after randomization
Number of patients requiring treatment with vasopressors | From date of randomization to 30 days
  Number of patients that die or number of patients that require treatment with vasopressors within 30 days after randomization

SECONDARY OUTCOMES:
Length of hospital stay | From date of randomization until date of documented hospital discharge or date of death from any cause, whichever came first, assessed up to 6 months
  Duration of hospital length of stay in days
Inhospital mortality | From date of randomization until date of death in hospital from any cause, assessed up to 6 months
  The number of death measured inhospital before discharge
30-days mortality | up to 30 days from baseline (randomization date)
  The number of death within 30 days
90-days mortality | Up to 90 days from baseline (randomization date)
  The number of death within 90 days
One-year mortality | Up to one-year from baseline (randomization date)
  The number of death within one-year
Five-year mortality | Up to five-years from baseline (randomization date)
  The number of death within five-years
Discharge within 24 hours | Up to 24 hours after rom baseline (randomization date)
  The number of patients discharged within 24 hours
Readmission | 30 days after discharge date
  The number of patients readmitted to hospital
Intensive care admission | From date of randomization until date of admission to intensive care during hospitalization due to any cause, assessed up to 6 months
  Number of patients admitted to intensive care during current hospital stay
Days on antibiotic treatment within 30 days | Within 30 days from randomization date
  Number of days the patient have been treated with antibiotics
Bacteremia | Day 7 to day 30 from randomization date
  Number of patients diagnosed with bacteremia

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No